CLINICAL TRIAL: NCT02646904
Title: Nebulized Beclometasone Dipropionate Improves Nasal Patency in Children With Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stefania La Grutta, MD (Other)
Responsible Party: Sponsor-Investigator, Stefania La Grutta, MD, MD, Senior Researcher, Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Organization: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9-2015
Record Dates: First submitted 2015-12-18; First posted 2016-01-06 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beclometasone Dipropionate (BDP) (Experimental): Standard dose (400 µg/daily as 100 µg 1 spray nos bid) of Nasal Beclomethasone Dipropionate for 21 days.
  Interventions: Drug: Nasal Beclomethasone Dipropionate
- CERCHIO 10 mg/ml OS (Active Comparator): For Children < 12 years old 10 drops die (5 mg die) for 21 days. For Children > 12 years old 20 drops die (10 mg die) for 21 days.
  Interventions: Drug: CERCHIO 10 mg/ml OS

INTERVENTIONS:
Drug: Nasal Beclomethasone Dipropionate — Standard dose (400 µg/daily as 100 µg 1 spray nos bid) of nebulized Beclomethasone Dipropionate nasal spray for 21 days.
  Other Names: NBDP
  Arms: Beclometasone Dipropionate (BDP)
Drug: CERCHIO 10 mg/ml OS — For Children < 12 years old 10 drops die (5 mg die) for 21 days. For Children > 12 years old 20 drops die (10 mg die) for 21 days.
  Arms: CERCHIO 10 mg/ml OS

SUMMARY:
The purpose of this study is to examine in children with persistent AR the effect of the topically applied beclomethasone in comparison with cetirizine on nasal patency evaluated by acoustic rhinometry and subjective nasal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* children 6-16 years of age with a history of AR in the previous year
* T5SS: ≥5 in the last week before enrollment

Exclusion Criteria:

* asthma symptoms
* acute upper respiratory infections
* anatomic nasal defects (ie, septum deviation), or nasal polyps
* use in the past 4 weeks of nasal or oral corticosteroids, nasal or oral decongestants, antihistamines.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Nasal patency evaluated by acoustic rhinometry. | 21 days
  The main objective is to assess the increase of nasal patency in children aged 6-16 with perennial allergic rhinitis (PAR), treated with Beclometasone nasal spray 100 µg/die for 21 days.

SECONDARY OUTCOMES:
Efficacy of Beclometasone nasal spray on subjective nasal symptoms | 21 days
  The secondary objective is to measure the impact of Beclometasone nasal spray 100 µg on subjective nasal symptoms, in children aged 6-16 with perennial allergic rhinitis (PAR), assessed by T4SS Questionnaire(Total 4 Symptoms Score).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Institute of Biomedicine and Molecular Immunology (IBIM), National Research Council, Palermo, Sicily
  - Institute of Biomedicine and Molecular Immunology, IBIM, Palermo

IPD SHARING:
Plan to Share IPD: Yes
The IPD collected will be available on February 2017.
  The following participant data will be shared:
  * Nasal patency
  * Nasal symptom score
  * Demographic characteristics
  All IPD will be obtained from statistical analysis on the dedicated database in which all data are stored.